CLINICAL TRIAL: NCT05408520
Title: A Randomized Controlled Trial of Targeted Muscle Reinnervation in Patients Requiring Lower Extremity Amputation.
Brief Title: Targeted Muscle Reinnervation Study (TMR)
Acronym: TMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Joshua Hustedt (Other)
Responsible Party: Sponsor-Investigator, Joshua Hustedt, Assistant Professor, Orthopedics, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000650
Record Dates: First submitted 2022-05-12; First posted 2022-06-07 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Amputation
Keywords: lower extremity amputation; neuroma; phantom limb pain; nerve damage; postoperative pain amputee; reinnervation; regenerative neurotization
MeSH Terms: conditions — Neuroma; Phantom Limb

STUDY DESIGN:
Intervention Model Description: A traditional amputation follows the normal standard of care, with transection of peripheral nerves. The TMR procedure will transfer the transected nerves to adjacent muscle nerves.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amputation with TMR (Experimental): Amputation will follow standard procedure, but with the addition of the TMR procedure, which involves rerouting severed or injured nerves to new muscle targets using microsurgical techniques to provide the nerve endings with a new muscle to innervate.
  Interventions: Procedure: Targeted Muscle Reinnervation
- Amputation without TMR (SOC) (No Intervention): A traditional amputation follows the normal standard of care, with transection of peripheral nerves.

INTERVENTIONS:
Procedure: Targeted Muscle Reinnervation — When a nerve is severed or injured, it attempts to regenerate. The TMR procedure will transfer the transected nerves to adjacent muscle nerves in efforts to encourage the nerve to regenerate in an organized fashion.
  Arms: Amputation with TMR

SUMMARY:
The purpose of this study is to examine the effect of targeted muscle reinnervation on the outcomes of amputees at a level 1 trauma center. The investigators propose to randomize all patients requiring amputation with and without targeted muscle reinnervation. This study will help delineate the efficacy of targeted muscle reinnervation in the general population.

DETAILED DESCRIPTION:
After an amputation, patients often experience pain, both from the cut nerves themselves as well as perceived pain from a 'missing' limb. A technique has been developed to regenerate the cut nerve so that it doesn't cause pain. The technique includes sewing the nerve into another nerve so that it continues to function. This technique, called targeted muscle reinnervation, can reduce the postoperative pain amputee patients experience.

Targeted muscle reinnervation (TMR) has shown promising success in the reduction of neuroma and phantom limb pain following extremity amputation. TMR was originally designed to allow for regenerative neurotization of end target muscle for the purpose of utilizing myoelectric prosthesis for amputees. While these indications have been successful, it has been the secondary outcome of reduction in neuroma and phantom limb pain that have led to significant improvements in patient outcomes.

In the United States there are 200,000 amputations every year, and 1.6 million Americans living as amputees. Despite the technical success of the procedures, over 75% of patients will experience neuroma pain, and 85% will experience phantom limb pain. In addition, this pain limits the postoperative ambulation of many patients leading to a 75% 5-year mortality rate for patients who undergo lower extremity amputation in the US.3 TMR has shown promising clinical results in addressing phantom limb and neuroma pain. In pooled data it showed that patients who underwent TMR had residual limb pain of 0% and phantom limb pain of 7%. In a larger comparative study of 489 patients, patients who underwent TMR had phantom limb pain scores with an average of 1, compared to an average of 5 for control amputees. The TMR patients also had an average residual limb pain of 1, compared to an average of 4 for controls.

Yet despite these promising outcomes, questions with TMR still remain. In the Valerio study, the largest study to date, all patients were grouped together regardless of the reason for amputation. While the percentage of patients undergoing amputation for cancer, infection, ischemia, trauma, or other, was reported, there was no comparison of outcomes in these groups. In a new study, the benefits of TMR have been shown to hold in highly comorbid patients presenting to a level 1 trauma center. Given the outcomes of TMR in these studies, there seems to be strong evidence to encourage the procedure, yet no study has yet to randomize patients to measure the true clinical outcome in a trauma population.

ELIGIBILITY:
Inclusion Criteria:

* Any individual 18 years and older indicated for a below knee or above knee amputation at Banner-University Medical Center Phoenix

Exclusion Criteria:

* Any individual who does not meet inclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Effect of TMR on neuroma | Pre-operative through 24 months
  Subject data will be collected from EMR and patient reported outcome surveys, rating pain on a scale of 1-10 (1 being no pain and 10 being the worst pain).
Effect of TMR on phantom limb pain | Pre-operative through 24 months
  Subject data will be collected from EMR and patient reported outcome surveys, rating pain on a scale of 1-10 (1 being no pain and 10 being the worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hustedt, MD, MHS, Principal Investigator — University of Arizona
Locations (1):
- Banner - University Medical Center, Phoenix campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Background] Bowen JB, Ruter D, Wee C, West J, Valerio IL. Targeted Muscle Reinnervation Technique in Below-Knee Amputation. Plast Reconstr Surg. 2019 Jan;143(1):309-312. doi: 10.1097/PRS.0000000000005133. PMID 30589808
- [Background] Kuiken TA, Dumanian GA, Lipschutz RD, Miller LA, Stubblefield KA. The use of targeted muscle reinnervation for improved myoelectric prosthesis control in a bilateral shoulder disarticulation amputee. Prosthet Orthot Int. 2004 Dec;28(3):245-53. doi: 10.3109/03093640409167756. PMID 15658637
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Bowen JB, Wee CE, Kalik J, Valerio IL. Targeted Muscle Reinnervation to Improve Pain, Prosthetic Tolerance, and Bioprosthetic Outcomes in the Amputee. Adv Wound Care (New Rochelle). 2017 Aug 1;6(8):261-267. doi: 10.1089/wound.2016.0717. PMID 28831329
- [Background] Souza JM, Cheesborough JE, Ko JH, Cho MS, Kuiken TA, Dumanian GA. Targeted muscle reinnervation: a novel approach to postamputation neuroma pain. Clin Orthop Relat Res. 2014 Oct;472(10):2984-90. doi: 10.1007/s11999-014-3528-7. PMID 24562875
- [Background] Valerio IL, Dumanian GA, Jordan SW, Mioton LM, Bowen JB, West JM, Porter K, Ko JH, Souza JM, Potter BK. Preemptive Treatment of Phantom and Residual Limb Pain with Targeted Muscle Reinnervation at the Time of Major Limb Amputation. J Am Coll Surg. 2019 Mar;228(3):217-226. doi: 10.1016/j.jamcollsurg.2018.12.015. Epub 2019 Jan 8. PMID 30634038
- [Background] Valerio I, Schulz SA, West J, Westenberg RF, Eberlin KR. Targeted Muscle Reinnervation Combined with a Vascularized Pedicled Regenerative Peripheral Nerve Interface. Plast Reconstr Surg Glob Open. 2020 Mar 25;8(3):e2689. doi: 10.1097/GOX.0000000000002689. eCollection 2020 Mar. PMID 32537346
- [Background] Dumanian GA, Potter BK, Mioton LM, Ko JH, Cheesborough JE, Souza JM, Ertl WJ, Tintle SM, Nanos GP, Valerio IL, Kuiken TA, Apkarian AV, Porter K, Jordan SW. Targeted Muscle Reinnervation Treats Neuroma and Phantom Pain in Major Limb Amputees: A Randomized Clinical Trial. Ann Surg. 2019 Aug;270(2):238-246. doi: 10.1097/SLA.0000000000003088. PMID 30371518
- [Background] Chang BL, Mondshine J, Attinger CE, Kleiber GM. Targeted Muscle Reinnervation Improves Pain and Ambulation Outcomes in Highly Comorbid Amputees. Plast Reconstr Surg. 2021 Aug 1;148(2):376-386. doi: 10.1097/PRS.0000000000008153. PMID 34398088